CLINICAL TRIAL: NCT01039636
Title: A PHASE 1b OPEN LABEL, MULTI-CENTER, ESCALATING MULTIPLE DOSE STUDY TO ASSESS THE SAFETY, TOLERABILITY, PHARMACOKINETICS AND PHARMACODYNAMICS OF FBS0701 IN PATIENTS WITH TRANSFUSIONAL IRON OVERLOAD
Brief Title: Safety and Pharmacokinetic Study of Escalating Multiple Doses of an Iron Chelator in Patients With Iron Overload
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FerroKin BioSciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FBS0701-CTP-03
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2011-01

CONDITIONS: Transfusional Iron Overload; Beta-thalassemia
Keywords: Beta-thalassemia; Sickle cell anemia; Transfusional iron overload; Iron overload; Iron chelation
MeSH Terms: conditions — beta-Thalassemia; Anemia, Sickle Cell; Iron Overload | interventions — 4,5-dihydro-2-(2-hydroxy-3-(3,6,9-trioxadecyloxy)phenyl)-4-methyl-4-thiazolecarboxylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FBS0701 - 5 escalating doses (Experimental): 5 escalating doses of FBS0701 in 5 cohorts of 4 patients each.
  Interventions: Drug: FBS0701

INTERVENTIONS:
Drug: FBS0701 — Oral FBS0701 for 7 days at one of the following doses: 3 mg/kg/day or 8 mg/kg/day or 16 mg/kg/day or 32 mg/kg/day or 40 mg/kg/day

SUMMARY:
The purpose of this research study is to study the safety of increasing doses of FBS0701, and to see how quickly the study medication is absorbed and how quickly it disappears from the bloodstream. FBS0701 is a new, oral iron chelator - a medication taken by mouth that increases the body's elimination of iron. Iron chelators are used in patients who develop iron overload from their transfusions. Four increasing doses of FBS0701 will be tested during this study. The study will start with the lowest dose given to 4 patients (3 mg/kg/day. The next group of 4 patients will receive the next high dose (8mg/kg/day only after the results of the first 4 patients are examined and it is determined safe to continue. Participating patients will take the study medication for 7 days and be followed for 28 days after their last dose to determine if they have any reactions to the study medication - therefore a total of 35 days on study. Patients will need to give up to 17 blood samples over the screening period and first 15 days of the study (a total of about 9 tablespoons). Patients will not need to stay overnight in the clinic but will need to visit the clinic 10 times for screening and on-study visits over the 35 days. Patients currently taking an iron chelator will need to stop that treatment for up to 22 days (up to 5 days before they start the study and for 15 days during the study). The results of this study will be helpful in determining the safety of the drug and the best doses of FBS0701 to be used in the next study which will assess the effectiveness of this new iron chelator.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Transfusion dependent (at least 8 transfusions per year) with transfusional iron overload needing treatment with deperoxamine, deferasirox or deperiprone.
* Willing to discontinue current iron chelation therapy for 2-5 days prior to enrollment and for a total of up to 3 weeks
* Willing to fast after midnight prior to each dose
* Serum ferritin greater than 400ng/ml
* Liver iron concentration greater than or equal to 1.5 mg iron. (determined by MRI or SQUID within 12 months prior to enrollment)
* Cardiac iron greater than or equal to 12 milliseconds (determined by MRI t2* within 18 months prior to enrollment)
* Mean of last 3 pre-transfusion hemoglobin values must be greater than or equal to 7.5 g/dl
* Agrees to use approved contraception from Screening and until 30 days after last administration of study drug. Abstinence OK.

Exclusion Criteria:

* Principal Investigator considers patient unfit for study after conducting a medical review, physical examination and other screening assessments.
* Non-elective hospitalization with past 30 days
* Evidence of clinically relevant oral, cardiovascular, gastrointestinal, hepatic, renal, endocrine, pulmonary, neurologic, psychiatric or skin disorder.
* Evidence of significant renal insufficiency; serum creatine above upper limit of normal or proteinuria greater than 2 gm per day or calculated creatinine clearance of less than or equal to 60ml/min
* Platelet count below 150,000,000/ml and/or absolute neutrophil count less then 1500/mm3
* Alkaline phosphatase or AST greater than 5 times the upper limit of normal or ALT greater than 4 times the upper limit of normal
* Female patients who are pregnant or lactating
* Use of any investigational agent within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability by AEs, Physical Exam, Clinical Laboratory assessments | 35 days (7 days treatment and 28 days follow up)
Steady state plasma level and half-life of FBS0701 | 7 days of dosing

SECONDARY OUTCOMES:
Urinary excretion of iron | 7 days of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Ellis Neufeld, MD, Principal Investigator — Boston Children's Hospital
Locations (5):
- United States (3):
  - Children's Hospital of Oakland, Oakland, California
  - Children's Hospital of Boston, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Royal Adelaide Hospital, Adelaide, Australia
- Siriraj Hospital, Mahidol University, Bangkok, Thailand